CLINICAL TRIAL: NCT00140140
Title: An Open-Label Phase I/II Study of Weekly ABI-007 and Vinorelbine With or Without G-CSF in Patients With Stage IV (Metastatic) Breast Cancer
Brief Title: A Phase I/II Study of ABI-007 (Abraxane®, Nab®-Paclitaxel)and Vinorelbine in Patients With Stage IV (Metastatic) Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to determine the optimum tolerated dose
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA025
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Stage IV (Metastatic) Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Vinorelbine; Trastuzumab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: 80 mg ABI-007 + 15 mg vinorelbine (Experimental): Weekly intravenous infusion of 80 mg/m^2 ABI-007, followed by an infusion of 15 mg/m^2 vinorelbine. Participants with human epidermal growth factor receptor 2-positive (HER2+) and who met cardiac safety requirements were also administered weekly Herceptin® (trastuzumab) following completion of ABI-007 and vinorelbine infusions. No G-CSF support was planned.
  Interventions: Drug: ABI-007; Drug: vinorelbine; Drug: Trastuzumab
- Part 2: 80 mg ABI-007 + 15 mg vinorelbine (Experimental): Weekly intravenous infusion of 80 mg/m^2 ABI-007, followed by an infusion of 15 mg/m^2 vinorelbine. Participants with human epidermal growth factor receptor 2-positive (HER2+) and who met cardiac safety requirements were also administered weekly Herceptin® (trastuzumab) following completion of ABI-007 and vinorelbine infusions. G-CSF support was given.
  Interventions: Drug: ABI-007; Drug: vinorelbine; Drug: Trastuzumab; Biological: G-CSF
- Part 2: 90 mg ABI-007 + 20 mg vinorelbine (Experimental): Weekly intravenous infusion of 90 mg/m^2 ABI-007, followed by an infusion of 20 mg/m^2 vinorelbine. Participants with human epidermal growth factor receptor 2-positive (HER2+) and who met cardiac safety requirements were also administered weekly Herceptin® (trastuzumab) following completion of ABI-007 and vinorelbine infusions. G-CSF support was given.
  Interventions: Drug: ABI-007; Drug: vinorelbine; Drug: Trastuzumab; Biological: G-CSF

INTERVENTIONS:
Drug: ABI-007 — Weekly intravenous infusions over 30 minutes.
  Other Names: Abraxane®; Nab®-Paclitaxel; paclitaxel protein-bound particles for injectable suspension
Drug: vinorelbine — Weekly intravenous infusions over 10-30 minutes, immediately after ABI-007. Vinorelbine is commercially available and was not supplied by the Sponsor.
  Other Names: Navelbine; vinorelbine tartrate; 5'noranhydrovinblastine
Drug: Trastuzumab — Trastuzumab was administered to participants who had HER-2-neu positive tumors. Participants received trastuzumab by IV infusion via a vascular access device following dosing with ABI-007 and vinorelbine. During their first cycle, 4 mg/kg was administered on day 1 of that cycle as a loading dose. During subsequent weekly treatments, 2 mg/kg was administered.
  Trastuzumab is commercially available and was not supplied by the Sponsor.
  Other Names: Herceptin
Biological: G-CSF — During Part 1, participants followed a dosing regimen with ABI-007 and vinorelbine without G-CSF treatment. However, G-CSF was allowed for administration as necessary in accordance with commonly accepted clinical guidelines.
  In Part 2, participants started G-CSF treatment in concurrence with their ABI-007 and vinorelbine treatments. G-CSF was administered to all participants on Days 2-7 of each cycle, at a dose of 5 mcg/kg. If the participant's absolute neutrophil (ANC) count was >20,000/mm^3 on the day of anticipated chemotherapy, the site staff reduced the daily dose of G-CSF by 50% to 2.5 mcg/kg.
  G-CSF is commercially available and was not supplied by the Sponsor.
  Other Names: granulocyte-colony stimulating factor
  Arms: Part 2: 80 mg ABI-007 + 15 mg vinorelbine; Part 2: 90 mg ABI-007 + 20 mg vinorelbine

SUMMARY:
The purpose of this study is to: 1) determine the optimal tolerated dose of ABI-007 and vinorelbine, given concurrently on a weekly basis, in the absence of planned growth factor support with granulocyte colony-stimulating factor (G-CSF) (Patients with HER-2/neu positive disease may receive Herceptin, and 2) determine the optimal tolerated dose of ABI-007 and vinorelbine, given concurrently on a weekly basis, in the presence of planned growth factor support with G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Patient has microscopically confirmed invasive breast carcinoma with clinical and/or radiographic evidence of stage 4 disease. If diagnosis is based on pleural effusion, positive cytology must be confirmed.
* Patient has had no prior chemotherapy for Stage 4 disease (hormone therapy is permitted). Prior adjuvant paclitaxel by 3-hour infusion is permitted, if there is no residual neuropathy. Prior adjuvant docetaxel on an every 3 week schedule is permitted.
* Disease must be measurable (unidimensional by Response Evaluation Criteria In Solid Tumors (RECIST) criteria) or evaluable (e.g., malignant effusion, marrow involvement). Elevated tumor markers alone are insufficient.
* Age >18.
* Southwest Oncology Group (SWOG)/Eastern Oncology Group (ECOG) performance status must be < or =2 at screen and on treatment day one.
* Life expectancy must be estimated at >16 weeks.
* Prior irradiation is permitted, provided:

  * Does not exceed 25% of the estimated bone marrow volume
  * Measurable/evaluable disease exists outside the radiation field, or progressive disease is documented within the radiation field.
* Informed consent must be obtained prior to registration.
* Patients must be > 2 weeks from prior surgery; > 3 weeks from radiation therapy to the pelvis, spine or long bones; > 3 weeks from prior chemotherapy (> 6 weeks for mitomycin C or nitrosureas), or > 2 weeks from prior hormonal therapy.
* All patients must have placement of appropriate central venous access device.
* Tumor HER2/neu expression must be determined prior to study enrollment. Assessment may be by fluorescence in situ hybridization (FISH) assay or by immunohistochemistry (ICC). If determination is intermediate by ICC, FISH must be performed. For enrollment purposes, this phase I study will not discriminate based on HER2 status. However, documentation of patients' HER2 status will be maintained and Herceptin will be prescribed for all HER2 positive patients.

Exclusion Criteria:

* Granulocytes < 1,500/mm^3.
* Platelets < 100,000/mm^3.
* Hemoglobin < 9 gm/dl.
* Creatinine > 2.0 mg/dl.
* Total bilirubin > 2 mg/dl.
* Visceral crisis characterized by rapidly progressive hepatic or lymphangitic lung metastases.
* Medically unstable as judged by the patient's physician.
* Pregnancy or lactation; failure to employ adequate contraception.
* Uncontrolled central nervous system (CNS) disease.
* Pre-existing Grade ≥ 2 peripheral neuropathy except for abnormalities due to cancer.
* Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol.
* Prior therapy with vinorelbine or prior therapy with a taxane that resulted in neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Care Center, Duarte, California
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Started | 4 | 6 | 6
Completed | 2 (Progressive disease) | 4 (Progressive disease) | 4 (Progressive disease)
Not Completed | 2 | 2 | 2
Not completed — Unacceptable toxicity | 1 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Customized [Number; unit: participants]
  < 65 years | 4 (5.74) | 5 (12.60) | 5 (12.23) | 14
  >= 65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 6 | 16
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 0 | 1
  White, Non-Hispanic and Non-Latino | 3 | 5 | 4 | 12
  White, Hispanic or Latino | 0 | 1 | 2 | 3
Menopausal Status [Number; unit: participants]
  Pre-menopausal | 1 | 2 | 1 | 4
  Post-menopausal | 3 | 4 | 5 | 12
Smoking Status [Number; unit: participants]
  Never Smoked | 2 | 4 | 3 | 9
  Current Smoker | 1 | 1 | 0 | 2
  Previous Smoker, but have Stopped | 1 | 1 | 3 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants]
  Status 0 (Asymptomatic) | 1 | 2 | 1 | 4
  Status 1 (Symptomatic but completely ambulatory) | 3 | 4 | 4 | 11
  Status 2 (Ambulatory but unable to work) | 0 | 0 | 1 | 1
  Status 3 (Limited self-care) | 0 | 0 | 0 | 0
  Status 4 (Completely disabled) | 0 | 0 | 0 | 0
  Status 5 (Death) | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Confirmed Complete or Partial Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0)
Description: Overall response rate (ORR) is complete response (CR) + partial response (PR). Complete response (CR): The disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation. All sites must be assessed, including non-measurable sites, such as effusions, or markers. Disappearance of all non-target lesions. The normalization of tumor marker level confirmed at least 4 weeks after initial documentation.
  Partial response (PR): At least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing. As well as persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Time Frame: up to month 30
Population: Treated population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
percentage of participants | 25 [0.6 to 80.6] | 16.7 [0.4 to 64.1] | 33.3 [4.3 to 77.7]

2. Primary Outcome: Participants With Dose Limiting Toxicities
Description: Toxicities were evaluated based on the U.S. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Any drug-related toxicities CTC Grade 3 or higher were considered dose limiting. Grade 3=severe AE, Grade 4=life-threatening or disabling AE, Grade 5=death. Other conditions considered dose-limiting toxicities include:
  * requirement of a dose adjustment during the first 4 weeks
  * a dose delay of >3 weeks during the first 4 weeks Grade 3 or greater toxicities attributed to the use of Herceptin were not considered dose-limiting toxicities.
  The optimal tolerated dose of ABI-007 and vinorelbine given concurrently was defined as the dose administered in the absence of DLTs.
Time Frame: up to month 1
Population: Treated population
Measure: Number; unit: participants
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
participants | 2 | 2 | 2

3. Primary Outcome: Percentage of Participants With Discontinued, Delayed or Interrupted Therapy
Description: Percentage of participants who had discontinued therapy or had a delayed dose or an interrupted (omitted) dose due to toxicities/adverse events.
Time Frame: up to week 129
Population: Treated population
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
percentage of participants
  At least 1 ABI-007 dose reduction | 50 | 50 | 17
  At least 1 Vinorelbine dose reduction | 50 | 50 | 17
  At least 1 ABI-007 dose interruption | 0 | 0 | 0
  At least 1 Vinorelbine dose interruption | 0 | 0 | 0
  At least 1 therapy delay | 75 | 83 | 67

4. Primary Outcome: Participant Counts of the Most Severe Grade for Absolute Neutrophil (ANC), White Blood Cell (WBC), Platelet, and Hemoglobin Counts as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Experience (NCI CTCAE v3)
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest measured (nadir) blood counts were graded using NCI CTCAE version 3.
  ANC:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 1.5*10^9/L; Grade 2 = <1.5 - 1.0*10^9/L; Grade 3 = <1.0 - 0.5*10^9/L; Grade 4 = <0.5*10^9/L
  WBC:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 3.0*10^9/L; Grade 2 = <3.0 - 2.0*10^9/L; Grade 3 = <2.0 - 1.0*10^9/L; Grade 4 = <1.0*10^9/L
  Platelets:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 75.0*10^9/L; Grade 2 = <75.0 - 50.0*10^9/L; Grade 3 = <50.0 - 25.0*10^9/L; Grade 4 = <25.0*10^9/L
  Hemoglobin:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 100 g/L ; Grade 2 = <100 - 80 g/L; Grade 3 = <80 - 65 g/L; Grade 4 = <65 g/L
Time Frame: up to week 129 (longest treatment)
Population: Treated population
Measure: Number; unit: participants
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
participants
  ANC: grade 0 | 1 | 1 | 3
  ANC: grade 1 | 1 | 1 | 0
  ANC: grade 2 | 0 | 1 | 0
  ANC: grade 3 | 2 | 0 | 1
  ANC: grade 4 | 0 | 3 | 2
  WBC: grade 0 | 2 | 3 | 1
  WBC: grade 1 | 0 | 0 | 1
  WBC: grade 2 | 1 | 1 | 2
  WBC: grade 3 | 1 | 2 | 2
  WBC: grade 4 | 0 | 0 | 0
  Platelets: grade 0 | 4 | 4 | 6
  Platelets: grade 1 | 0 | 1 | 0
  Platelets: grade 2 | 0 | 1 | 0
  Platelets: grade 3 | 0 | 0 | 0
  Platelets: grade 4 | 0 | 0 | 0
  Hemoglobin: grade 0 | 0 | 1 | 0
  Hemoglobin: grade 1 | 2 | 0 | 0
  Hemoglobin: grade 2 | 1 | 3 | 4
  Hemoglobin: grade 3 | 1 | 2 | 2
  Hemoglobin: grade 4 | 0 | 0 | 0

5. Primary Outcome: Nadir Measurement for Absolute Neutrophil (ANC), White Blood Cell (WBC) and Platelet Count
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest observed measurement is the nadir. Blood counts were performed each week of treatment.
Time Frame: up to week 129 (longest treatment)
Population: Treated population
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
10^9/L
  ANC | 1.74 (1.444) | 1.00 (0.864) | 1.72 (1.589)
  WBC | 2.79 (0.999) | 2.56 (0.962) | 2.92 (1.572)
  Platelets | 221.5 (108.19) | 187.2 (70.35) | 222.7 (50.11)

6. Primary Outcome: Nadir Measurement for Hemoglobin (Hgb)
Description: as for outcome 5
Time Frame: up to week 129 (longest treatment)
Population: Treated population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
g/L | 89.3 (16.11) | 89.7 (14.53) | 83.5 (6.09)

7. Secondary Outcome: Percentage of Participants With Stable Disease for >= 16 Weeks, or Complete or Partial Response According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0)
Description: Disease control is stable disease (SD) for >=16 weeks + complete response (CR) + partial response (PR). See Outcome #1 for definitions of CR and PR.
  RECIST defines SD for target lesions as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: up to month 30
Population: Treated population
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
percentage of participants
  Disease control | 75 | 66.7 | 33.3
  Complete response | 0 | 0 | 0
  Partial response | 25 | 17 | 33
  Stable disease >=16 weeks | 50 | 50 | 0

8. Secondary Outcome: Kaplan Meier Estimate for Time to Disease Progression (TTP)
Description: Time to progression was defined as the time from the first dose of study drug to the start of progression. Participants that did not have progression were censored at the last known time the patient was evaluated for progression. Participants that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: up to month 30
Population: Treated population of participants with disease progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 3 | 5 | 4
months | 8.8 [1.0 to 30.4] | 7.9 [3.5 to 16.4] | 4.2 [3.5 to 14.5]

9. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response
Description: Duration of response is defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or patient death from any cause, whichever occurred first. Patients that did not have progression or have not died were censored at the last known time the patient was progression free. Patients that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Complete response (CR) and partial response (PR) are defined in outcome #1. Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: up to month 30
Population: Treated participants who had a response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 1 | 1 | 2
months | 10.4 | 7.9 | 9.6 [4.6 to 14.5]

10. Secondary Outcome: Kaplan Meier Estimate for Progression-Free Survival (PFS)
Description: PFS was defined as the time from the first dose of study drug to the start of progression or patient death (any cause) whichever occurred first. Participants that did not have progression or have not died were censored at the last known time the participant was progression free. Participants that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Because no patients died as a result of a non-disease progression event, the analysis of PFS was identical to the analysis for TTP.
Time Frame: up to month 30
Population: Treated population of participants who had disease progression or who died
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 3 | 5 | 4
months | 8.8 [1.0 to 30.4] | 7.9 [3.5 to 16.4] | 4.2 [3.5 to 14.5]

11. Secondary Outcome: Kaplan-Meier Estimates for Participant Survival
Description: Participant survival is the time from the first dose of study drug to participant death from any cause. Participants that did not die were censored at the last known time the participant was alive.
Time Frame: up to 39 months
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 80 mg ABI-007 + 15 mg Vinorelbine | Part 2: 90 mg ABI-007 + 20 mg Vinorelbine
Number analyzed (Participants) | 4 | 6 | 6
months | 32.7 [3.1 to 32.7] | 29.2 [25.2 to 29.2] | 22.2 [19.4 to 26.1]

ADVERSE EVENTS:
Time Frame: Day 1 - up to 133 weeks (longest treatment plus 4 weeks)
Groups:
- 80 mg ABI-007 + 15 mg Vinorelbine: Weekly intravenous infusion of 80 mg/m^2 ABI-007, followed by an infusion of 15 mg/m^2 vinorelbine. Participants from study Parts 1 and 2 are combined.
- 90 mg ABI-007 + 20 mg Vinorelbine: Weekly intravenous infusion of 90 mg/m^2 ABI-007, followed by an infusion of 20 mg/m^2 vinorelbine. Participants are from study Part 2.
Arm/Group | 80 mg ABI-007 + 15 mg Vinorelbine | 90 mg ABI-007 + 20 mg Vinorelbine
Serious Adverse Events (participants affected / at risk) | 5/10 | 1/6
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 80 mg ABI-007 + 15 mg Vinorelbine (N=10) | 90 mg ABI-007 + 20 mg Vinorelbine (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 80 mg ABI-007 + 15 mg Vinorelbine (N=10) | 90 mg ABI-007 + 20 mg Vinorelbine (N=6)
Anemia (Blood and lymphatic system disorders) | 8 | 6
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 3 | 0
Lacrimation increased (Eye disorders) | 4 | 1
Vision blurred (Eye disorders) | 2 | 0
Visual acuity reduced (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0
Post procedural nausea (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Catheter related complication (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 0 | 1
Catheter site rash (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 8 | 5
Gait abnormal (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema mucosal (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 4 | 1
Pyrexia (General disorders) | 4 | 2
Rigors (General disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Blister (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Hepatic trauma (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3
Aspartate aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 4
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 4
Blood calcium decreased (Investigations) | 2 | 1
Blood chloride increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Haematocrit (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 3 | 1
Iron binding capacity total decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 6 | 2
Platelet count decreased (Investigations) | 2 | 0
Protein total decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 8 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Facial pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Lymphoedema (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Celgene shall complete its review within 30 days after receipt of a proposed publication or presentation submitted by the investigator. Upon request, the publication/presentation might be delayed up to 60 additional days for Celgene to secure intellectual property protection. Subsequent to the multicenter publication or one year after study completion, whichever occurs first, an investigator and/or his/her colleagues may publish the results of INVESTIGATOR's part of the study independently.